CLINICAL TRIAL: NCT01942642
Title: Evaluation of Dry Eye and Meibomian Gland Dysfunction After Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0690
Record Dates: First submitted 2013-08-29; First posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Meibomian Gland Dysfunction
Keywords: cataract surgery, meibomian gland dysfunction, meibum expressibility, meibography
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Meibomian gland dysfunction (MGD) is a common and important disease has been investigated the pathophysiology, diagnosis, treatment modalities of MGD, however, the changes of MGD after the cataract surgery, the most popular surgery to ophthalmologist, had not been evaluated. The investigators evaluated parameters related with MGD including lid margin abnormalities, meibomian gland expressibility and meibography before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for cataract surgery

Exclusion Criteria:

1. other comorbid ocular diseases such as ocular allergies.
2. continuous use of topical ocular medications before surgery
3. histories of ocular surgery, or ocular injury
4. Already had severe obstructive MGD before surgery, abnormal findings on lid margin (> 3 positive findings), reduced meibum expression (> grade 2), and obstructed gland dropout (meibography score > 3)

Ages: 45 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cataract surgery
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Ocular parameters | change of Ocular parameters from 1 to 3 months after cataract surgery
  Ocular symptom score, lid margin abnormalities, superficial punctuate keratopathy, tear film break-up time, Shirmer's test, lower tear meniscus height (TMH), depth (TMD), and area (TMA), meibum expressibility, and meibography score